CLINICAL TRIAL: NCT06223594
Title: Evaluation of Intravenous Fluid Therapy Within Dallas Acute Pancreatitis Protocol
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 028.PHA.2023.D
Record Dates: First submitted 2023-11-13; First posted 2024-01-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-07

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Intravenous Fluid Therapy — Evaluate the safety and efficacy of the Dallas acute pancreatitis protocol(DAPP) order set on Acute pancreatitis(AP) patients receiving aggressive, goal-directed Intravenous fluid(IVF )therapy.

SUMMARY:
Acute pancreatitis (AP) is a common disease of the gastrointestinal tract that can result in emotional, physical, and financial burdens on the patient.

DETAILED DESCRIPTION:
In the last 20 years, the incidence of AP and rate of hospitalization have steadily increased. Approximately, two-thirds of AP patients will have a mild and self-limiting course of the disease, leaving the remaining one-third experiencing moderately severe to severe disease that is associated with worse outcomes. Overall, the estimated mortality of pancreatitis is 1% however, mortality can be as high as 30% to 40% among patients with AP and organ failure or pancreatic necrosis. Despite numerous randomized clinical trials, there is no medication shown to be successful at treating AP.

AP is associated with fluid deficit secondary to low intake and vomiting. Early intravenous fluid (IVF) resuscitation has been long-established as the initial cornerstone treatment to prevent hypovolemia and subsequent organ failure within the first 48 to 72 hours. The rationale for such intervention is to provide adequate intravascular volume support to counteract fluid shift into the third space. However, available evidence for an effective fluid regimen is lacking with regard to the type of fluid, the optimal rate of administration, and how to assess appropriate goals/targets for adequate resuscitation. Furthermore, the literature has presented conflicting results on whether aggressive versus goal-directed fluid resuscitation will lead to a reduction in mortality and improve outcomes. Although early supportive care with IVF therapy is recommended by the major guidelines, there are potential, serious complications associated with aggressive resuscitation, including volume overload, respiratory failures, intra-abdominal compartments.

ELIGIBILITY:
Inclusion Criteria:

* ● Age > 18 years

  * Diagnosis of AP based on International Statistical Classification of Diseases( ICD)-10 code

Exclusion Criteria:

* ● Diagnosis of chronic pancreatitis

  * Patients who did not follow the IVF infusion protocol
  * Received < 24 hours of IVF therapy
  * Transferred from another institution

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Age > 18 years
  * Diagnosis of AP based on ICD-10 code
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Rate of fluid overload | 72 hours
  Rate of fluid overload at 72 hours, which is the absence of acute respiratory distress syndrome.

SECONDARY OUTCOMES:
number of Effective outcomes | 48 hours
  decrease in number days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Crotty, PharmD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI is committed to disseminate research results in a timely fashion. Sharing of data generated by this project will be carried out through presentation at scientific meetings and/or publication in Open Access Journals
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years